CLINICAL TRIAL: NCT03223025
Title: Efficacy and Safety of CinnaGen Recombinant Human Growth Hormone (CinnaTropin®) in Comparison With Novo Nordisk Growth Hormone (Nordilet®) Product in Pre-Pubertal Children With Idiopathic Growth Hormone Deficiency (IGHD)
Brief Title: Comparing Efficacy and Safety of CinnaGen Biosimilar Growth Hormone (CinnaTropin®) Versus Nordilet in Children With Idiopathic Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GH.CIN.MR93; IRCT201409064920N5 (Registry Identifier: Food And Drug Administration of The Islamic Republic of Iran)
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Idiopathic Growth Hormone Deficiency
Keywords: IGHD; somatropin
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CinnaTropin®, Then Nordilet® (Experimental): CinnaTropin® was administered with 0.03 mg/kg daily subcutaneous injections for three months. After that, the participants received 0.03 mg/kg daily subcutaneous injections of Nordilet® for three months.
  Interventions: Drug: CinnaTropin®; Drug: Nordilet®
- Nordilet®, Then CinnaTropin® (Active Comparator): Nordilet® was administered with 0.03 mg/kg daily subcutaneous injections for three months. After that, the participants received 0.03 mg/kg daily subcutaneous injections of CinnaTropin® for three months.
  Interventions: Drug: CinnaTropin®; Drug: Nordilet®

INTERVENTIONS:
Drug: CinnaTropin® — 0.03 mg/kg daily subcutaneous injections
  Other Names: recombinant human growth hormone (CinnaTropin®)
Drug: Nordilet® — 0.03 mg/kg daily subcutaneous injections
  Other Names: recombinant human growth hormone (Nordilet®)

SUMMARY:
This randomized, active-controlled, two-armed, open-label, and cross-over trial was designed to compare efficacy and safety of 0.03 mg/kg/day subcutaneous injections of either CinnaTropin® or Novo Nordisk growth hormone product in 30 children with Idiopathic Growth Hormone Deficiency. Patients were randomized to receive one of the products for three months. After that, each patient crossed over to the other arm to receive the other product for another three months. The primary objective of this study was to compare the efficacy of CinnaGen growth hormone (GH) with Nordilet. The secondary objectives of this study were further comparison and evaluation of efficacy along with safety between CinnaTropin® and Nordilet®.

DETAILED DESCRIPTION:
This study was a national, single center, randomized, active-controlled, two-arm, cross-over clinical trial to compare efficacy and safety of CinnaTropin® with Novo Nordisk growth hormone product in children with Idiopathic Growth Hormone Deficiency (IGHD).

After signing the written informed consent, patients were randomized to receive daily subcutaneous injections of CinnaTropin® or reference product (0.03mg/kg/day). Patients were admitted to receive the medication based on planned treatment. After three months patients were switched to receive the other product for another three months. Treatment visits were monthly for both groups.

The primary objective of this study is to compare the efficacy of CinnaTropin® with Novo Nordisk growth hormone product. The secondary objectives of this study are to further evaluation efficacy and safety.

During the trial, if patients bone age reached 14 and the improvement in their height was less than 2.5 cm than last year or, they did not reach the desired height appropriate for their age and gender or, if the growth plates were closed and they couldn't reach appropriate adulthood height, treatment will be discontinued.

The clinical trial was according to procedures that incorporate the ethical principles of GCP. Accurate and reliable data collection was assured by verification and cross-check of the CRFs against the patient's records by clinical monitors (source document verification was performed), and the maintenance of a drug-dispensing log by the center. A comprehensive validation check program was used to verify the data, and discrepancy reports were generated accordingly for resolution by the investigator.

Determination of sample size was based on the mean growth velocity of 9.7±1.3 following treatment with growth hormone and under consideration of 80% power, a sample size of 6 patient in each group was calculated. By considering patient loss and in order to increase the statistical power of the study a sample size of 15 patients in each group was determined.

ELIGIBILITY:
Inclusion Criteria:

* • Pre-pubertal boys and girls between 4-16 years (Tanner's stage 1)

  * Height Standard Deviation Score (HSDS) ≤ -2 SD for chronological age (Brandt/Reinken)
  * Approved GH Deficiency following clonidine GH stimulation test (150 µg/ m2, up to a maximum of 0.2 mg), and determining GH levels at 0, 30, 60, 90, and 120 minutes. This test is performed by overnight fasting and considered positive if GH ≥ 10 ng/ml, otherwise GHD is relevant.
  * Ruling out of other causes of short stature (hypothyroidism, Celiac disease, and etc.)
  * Documented Pituitary or hypothalamic hormone deficiency and below normal serum IGF-1 at the time of diagnosis
  * In case of the deficiency in other pituitary hormones, the patient can only be included, if the replacement of other pituitary hormones was done, and this is determined by the replacement of glucocorticoids provided that no symptoms of Cushing's syndrome be present, and the replacement of thyroxine and reaching to normal levels of free T4 and free T3.

Exclusion Criteria:

* • Any Illness that prevent the proper conduct of the trial, such as seizure, acute or systemic infectious disease in the past 6 months, chronic pulmonary infection, AIDS, chronic liver disease (verified disease of the hepatic cells or 2-fold or more increase in liver enzymes)

  * Any active malignancy (such as leukemia, etc.),
  * Contraindications of the administration of growth hormone (sleep apnea syndrome)
  * Turner syndrome.
  * Short stature due to chronic renal failure, other causes of GHD, such as craniopharyngioma
  * History of diabetes in patient or his/her first-degree relatives
  * Concomitant use of steroids

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2017-02-04 (Actual); Study Completion 2017-02-04 (Actual)

PRIMARY OUTCOMES:
Height velocity | three months
  The primary outcome of this study is to compare height velocity of patients in each treatment arm. Height velocity is reported in terms of centimeters per year.

SECONDARY OUTCOMES:
Height | three months
  Changes in height is measured in both treatment arms.
Weight | three months
  Changes in height is measured in both treatment arms.
Bone Age | six months
  Bone age is determined by wrist x-ray radiography in both treatment arms
HSDS | three months
  Height standard deviation score is calculated to compare height based on reference population.
HVSDS | three months
  Height velocity standard deviation score (HVSDS) is calculated to assess height velocity based on reference population.
The incidence of Adverse Events | three months; From receiving the first dose of each recombinant human growth hormone product until the last dose;
  The incidence of adverse events at each visit is recorded based on patients' reports, vital signs, physical examinations, and laboratory tests for systemic safety, including liver function, renal function, complete blood count and clinical chemistries, urinalysis, and hematologic testing.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kato Y, Murakami Y, Sohmiya M, Nishiki M. Regulation of human growth hormone secretion and its disorders. Intern Med. 2002 Jan;41(1):7-13. doi: 10.2169/internalmedicine.41.7. PMID 11838603
- [Background] Henwood MJ, Grimberg A, Moshang T Jr. Expanded spectrum of recombinant human growth hormone therapy. Curr Opin Pediatr. 2002 Aug;14(4):437-42. doi: 10.1097/00008480-200208000-00015. PMID 12130909
- [Background] Frindik JP, Kemp SF, Sy JP. Effects of recombinant human growth hormone on height and skeletal maturation in growth hormone-deficient children with and without severe pretreatment bone age delay. Horm Res. 1999;51(1):15-9. doi: 10.1159/000023307. PMID 10095164
- [Background] Lanes R. Growth velocity, final height and bone mineral metabolism of short children treated long term with growth hormone. Curr Pharm Biotechnol. 2000 Jul;1(1):33-46. doi: 10.2174/1389201003378997. PMID 11467359
- [Background] Shulman DI, Root AW, Diamond FB, Bercu BB, Martinez R, Boucek RJ Jr. Effects of one year of recombinant human growth hormone (GH) therapy on cardiac mass and function in children with classical GH deficiency. J Clin Endocrinol Metab. 2003 Sep;88(9):4095-9. doi: 10.1210/jc.2003-030030. PMID 12970269
- [Background] Bernasconi S, Arrigo T, Wasniewsk M, Ghizzoni L, Ruggeri C, Di Pasquale G, Vottero A, De Luca F. Long-term results with growth hormone therapy in idiopathic hypopituitarism. Horm Res. 2000;53 Suppl 1:55-9. doi: 10.1159/000053206. PMID 10895044
- [Background] Gasperi M, Aimaretti G, Scarcello G, Corneli G, Cosci C, Arvat E, Martino E, Ghigo E. Low dose hexarelin and growth hormone (GH)-releasing hormone as a diagnostic tool for the diagnosis of GH deficiency in adults: comparison with insulin-induced hypoglycemia test. J Clin Endocrinol Metab. 1999 Aug;84(8):2633-7. doi: 10.1210/jcem.84.8.5904. PMID 10443652
- [Background] Biller BM, Vance ML, Kleinberg DL, Cook DM, Gordon T. Clinical and reimbursement issues in growth hormone use in adults. Am J Manag Care. 2000 Sep;6(15 Suppl):S817-27. PMID 11184423
- [Background] Bright GM, Julius JR, Lima J, Blethen SL. Growth hormone stimulation test results as predictors of recombinant human growth hormone treatment outcomes: preliminary analysis of the national cooperative growth study database. Pediatrics. 1999 Oct;104(4 Pt 2):1028-31. PMID 10506258
- [Background] Janssen YJ, Frolich M, Roelfsema F. The absorption profile and availability of a physiological subcutaneously administered dose of recombinant human growth hormone (GH) in adults with GH deficiency. Br J Clin Pharmacol. 1999 Mar;47(3):273-8. doi: 10.1046/j.1365-2125.1999.00892.x. PMID 10215751
- [Background] Drake WM, Howell SJ, Monson JP, Shalet SM. Optimizing gh therapy in adults and children. Endocr Rev. 2001 Aug;22(4):425-50. doi: 10.1210/edrv.22.4.0438. PMID 11493578
- [Background] De Muinck Keizer-Schrama S, Rikken B, Hokken-Koelega A, Wit JM, Drop S. Comparative effect of two doses of growth hormone for growth hormone deficiency. The Dutch Growth Hormone Working Group. Arch Dis Child. 1994 Jul;71(1):12-8. doi: 10.1136/adc.71.1.12. PMID 8067786
- [Background] Soliman AT, abdul Khadir MM. Growth parameters and predictors of growth in short children with and without growth hormone (GH) deficiency treated with human GH: a randomized controlled study. J Trop Pediatr. 1996 Oct;42(5):281-6. doi: 10.1093/tropej/42.5.281. PMID 8936959
- [Background] Rikken B, van Doorn J, Ringeling A, Van den Brande JL, Massa G, Wit JM. Plasma levels of insulin-like growth factor (IGF)-I, IGF-II and IGF-binding protein-3 in the evaluation of childhood growth hormone deficiency. Horm Res. 1998 Sep;50(3):166-76. doi: 10.1159/000023268. PMID 9762006